CLINICAL TRIAL: NCT05253950
Title: The Effect of Technology on the Occurrence of Muscoskeletal Disorders in Students of A&B
Brief Title: Technology on the Occurrence of Muscoskeletal Disorders in Students
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Konstantinos Chandolias, Adjunct Lecturer, Member of Health Assessment and Quality of life Research Labοratory, clinical researcher, University of Thessaly
Other Study IDs: KC26042015
Record Dates: First submitted 2022-01-20; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Pain, Chronic; Posture Disorders in Children
Keywords: musculetical pain; electronic device; addiction; posture
MeSH Terms: conditions — Chronic Pain; Behavior, Addictive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Group: A sample of 120 people was collected from all over Greece, more specifically 7.6% belong to the region of Attica, 7.6% belong to the region of Western Greece, 0.8% belong to the region of Thessaly, 32.8% belong to the region of Central Macedonia and 51.3% belong to the region of Crete .
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — answered questions from two standard questionnaires the Internet Addiction Test (IAT) which examines students' dependence on the internet and the Nordic Muscuskeletal Questionnaire (NQS) which examines the onset of symptoms from the musculoskeletal system

SUMMARY:
To investgate the long use of electronic devices that forces the person to adopt an uncomfortable posture which leads to the appearance of musculoskeletal disorders such as neck pain, thoracic pain, back pain and tendonitis of the upper extremities due to writing messages and especially when the person uses only one hand.

DETAILED DESCRIPTION:
Due to the uncontrolled use of electronic devices, the purpose of this research is to initially prove that the long-term use of electronic devices is a factor in the occurrence of pain in the musculoskeletal system in students of A '& B' of High school. A secondary question of the present study is the hypothesis that adopting the wrong posture while using smart devices plays an important role in the onset of symptoms in one or more parts of the body. Finally, the third research question of the present study concerns whether long-term use of electronic devices is responsible for reducing physical activity in students.

In order to prove the positive correlation between technology and musculoskeletal disorders but also to answer the above questions, a questionnaire was distributed online to one hundred and twenty students of A '& B' Lyceum from all over Greece, which was promoted online. More specifically, the questionnaire included questions from two standard questionnaires, the Internet Addiction Test (IAT) and the Nordic Muscuskeletal Questionnaire (NQS).In addition they completed a medical history and supplementary questions about their physical condition and the attitudes they adopt when using electronic devices.

ELIGIBILITY:
Inclusion Criteria:

* without psychiatric disorders
* attended the A & B High School

Exclusion Criteria:

* undergone surgery on the musculoskeletal system

Ages: 15 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: A sample of 120 people was collected from all over Greece, more specifically 7.6% belong to the region of Attica, 7.6% belong to the region of Western Greece, 0.8% belong to the region of Thessaly, 32.8% belong to the region of Central Macedonia and 51.3% belong to the region of Crete . Criteria for participation in the research were students who were competent, without psychiatric disorders who attended the A & B High School, while the exclusion criteria from the research were students who have undergone surgery on the musculoskeletal system.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Nordic Musculoskeletal Questionnaire (NQS) | 1 day
  Long-term use of electronic devices in the occurrence of musculoskeletal disorders on neck pain, on shoulder pain, on hip pain, on knees pain, on fingers pain
Internet Addiction Test (IAT) | 1 day
  Incorrect posture and long use of electronic devices as a cause of musculoskeletal disorders, during the use of the mobile phone in a sitting position, in lying down and in standing position.
Internet Addiction Test (IAT) | 1 day
  Low physical condition and long use of electronic devices
Nordic Musculoskeletal Questionnaire (NGS) | 1 day
  Investigation of pain treatment of students who reported symptoms in the musculoskeletal system by medical help or medication to treat pain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Thessaly, Lamía, Central Macedonia, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Wolf, C., Wolf, S., Weiss, M., & Nino, G. (2018). Children's environmental health in the digital era: understanding early screen exposure as a preventable risk factor for obesity and sleep disorders. Children, 5(2), 31. 2. Canillas, F., Colino, A., & Menéndez, P. (2014). Cellular phone overuse as a cause for trapeziometacarpal osteoarthritis: a two case report. Journal of orthopaedic case reports, 4(4), 6. 3. Kim, H. J., & Kim, J. S. (2015). The relationship between smartphone use and subjective musculoskeletal symptoms and university students. Journal of physicaltherapyscience, 27(3), 575-579. 4. Eitivipart, A. C., Viriyarojanakul, S., & Redhead, L. (2018). Musculoskeletal disorder and pain associated with smartphone use: A systematic review of biomechanical evidence. Hong Kong Physiotherapy Journal, 38(02), 77-90. 5. Lepp, A., Barkley, J. E., Sanders, G. J., Rebold, M., & Gates, P. (2013). The relationship between cell phone use, physical and sedentary activity, and cardiorespiratory fitness in a sample of US college students. International Journal of Behavioral Nutrition and physical activity, 10(1), 1-9 6. Billieux, J., Philippot, P., Schmid, C., Maurage, P., De Mol, J., & Van der Linden, M. (2015). Is dysfunctional use of the mobile phone a behavioural addiction? confronting symptom-based versus process-based approaches. Clinical psychology & psychotherapy, 22(5), 460-468. 7. Jung, S. I., Lee, N. K., Kang, K. W., Kim, K., & Do, Y. L. (2016). The effect of smartphone usage time on posture and respiratory function. Journal of physical therapy science, 28(1), 186-189. 8. Knapik, J. J. (2015). The importance of physical fitness for injury prevention: part 1. Journal of special operations medicine: a peer reviewed journal for SOF medical professionals, 15(1), 123-127. 9. Penglee, N., Christiana, R. W., Battista, R. A., & Rosenberg, E. (2019). Smartphone use and physical activity among college students in health science-related majors in the United States and Thailand. International journal of environmental research and public health, 16(8), 1315. 10. Gustafsson, E. (2012). Ergonomic recommendations when texting on mobile phones. Work, 41(Supplement 1), 5705-5706. 11. Cramer, H., Mehling, W. E., Saha, F. J., Dobos, G., & Lauche, R. (2018). Postural awareness and its relation to pain: validation of an innovative instrument measuring awareness of body posture in patients with chronic pain. BMC musculoskeletal disorders, 19(1), 1-10. 12. Brumagne, S., Janssens, L., Janssens, E., & Goddyn, L. (2008). Altered postural control in anticipation of postural instability in persons with recurrent low back pain. Gait & posture, 28(4), 657-662. 13. Revel, M., Andre-Deshays, C., & Minguet, M. (1991). Cervicocephalic kinesthetic sensibility in patients with cervical pain. Archives of physical medicine and rehabilitation, 72(5), 288-291. 14. Brumagne, S., Cordo, P., Lysens, R., Verschueren, S., & Swinnen, S. (2000). The role of paraspinal muscle spindles in lumbosacral position sense in individuals with and without low back pain. Spine, 25(8), 989-994. 15. Langford, M. L. (1994). Poor posture subjects a worker's body to muscle imbalance, nerve compression. Occupational Health & Safety (Waco, Tex.), 63(9), 38-40. 16. Borhany, T., Shahid, E., Siddique, W. A., & Ali, H. (2018). Musculoskeletal problems in frequent computer and internet users. Journal of family medicine and primary care, 7(2), 337. 17. Ellahi, A., Khalil, M. S., & Akram, F. (2011). Computer users at risk: Health disorders associated with prolonged computer use. Journal of Business Management and Economics, 2(4), 171-182.